CLINICAL TRIAL: NCT05445011
Title: Safety and Efficacy of Anti-FLT3 CAR- T Cell (TAA05 Cell Injection) in the Treatment of Relapsed/ Refractory Acute Myeloid Leukemia
Brief Title: Anti-FLT3 CAR-T Cell (TAA05 Cell Injection) in the Treatment of Relapsed / Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, MEI HENG, Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti-FLT3 CAR-T Cell
Record Dates: First submitted 2022-06-23; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: FLT3 positive Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAA05 Cell Injection (Experimental): Fludarabine + Cyclophosphamide + TAA05 Cell Injection Patients will receive lymphodepletion with fludarabine (25 mg/kg) and cyclophosphamide (250 mg/kg) for 3 days on day -7~-2, followed by the infusion of TAA05 Cell with the dose of 1×10^8, 2×10^8 or 4×10^8 cells on day 0. If no dose-limited toxicity(DLT) emerges in the group, then the subsequent higher dose will be used in the next group. If DLT emerges in a single subject in any dose level, 3 more subjects will be enrolled to the same dose level. After the end of dose climbing, if the maximum dose group(MTD) is still not observed, the highest dose group is defined as MTD.
  Interventions: Drug: Fludarabine + Cyclophosphamide + TAA05 Cell Injection

INTERVENTIONS:
Drug: Fludarabine + Cyclophosphamide + TAA05 Cell Injection — Fludarabine + Cyclophosphamide + TAA05 Cell Injection Fludarabine 25 mg/kg * 3d on day-7~-2; Cyclophosphamide 250 mg/kg *3d on day-7~-2; TAA05 Cell Injection on day 0.
  Other Names: Fludarabine + Cyclophosphamide + Anti-FLT3 CAR-T Cell

SUMMARY:
This is a clinical trial of Anti-FLT3 CAR-T Cell (TAA05 Cell Injection) in the treatment of patients with relapsed / refractory acute myeloid leukemia. The purpose is to evaluate the safety and efficacy of anti-FLT3 CAR-T cells in patients with relapsed / refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a hematological malignancy characterized by clonal proliferation of hematopoietic stem cells or progenitor cells. AML is the most common type of leukemia in adults; the 5-year survival rate is only 24%. Moreover, 40%-50% of young patients and most elderly patients eventually suffered relapses.

FMS-like tyrosine kinase 3 (FLT3) is a member of the class III receptor tyrosine kinases, mainly expressed on the cell surface of hematopoietic progenitor cells and plays an important role in normal hematopoiesis such as proliferation, differentiation and survival. The variable expression of FLT3 can be found on leukemia blasts from over 90% of AML patients. Although about 30% of AML have FLT3 gene mutations, the ectodomain of the FLT3 molecule is usually spared so that cellular immunotherapy against it has great therapeutic potential. It is shown that FLT3 expression is detected in more than half of hematopoietic stem cell (HSC) and multipotent progenitor (MPP) cells on average, while the average positive rate of lymphoid progenitor (CLP) cells is less than 20%. Since the expression level of FLT3 on hematopoietic cells is not as high as CD33 and CD123, potential hematological toxicity has been supposed to be less obstructive to the development of FLT3-CAR-T Cell products. Besides, the expression of FLT3 is not found in other normal tissues. And it is reported that FLT3 CAR T cells did not deplete CD34(+) HSCs and preserve HSC differentiation in the mice model. Therefore, conducting CAR-T cell therapy targeting the FLT3 molecule could be very promising in the clinical practice of treating AML. TAA05 Cell Injection is a kind of FLT3-targeted CAR-T cell containing an optimized CD28 costimulatory domain which could help reduce the risk of toxic side effects. This clinical trial aims to evaluate the safety and efficacy of TAA05 Cell Injection in patients with FLT3 positive AML.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 ~ 70 years old (including boundary value), regardless of gender;
2. FLT-3 positive acute myeloid leukemia;
3. The expected survival time was more than 3 months;
4. ECOG score 0-2;
5. Refractory or relapsed AML patients after standardized treatment who meet any of the following criteria:

   1. After complete remission (CR), there were ≥5% leukemia cells or blast cells in the bone marrow(except for other reasons such as bone marrow regeneration after consolidation chemotherapy)in the peripheral blood and extramedullary lesions;
   2. Naive patients who are treated with 2 courses of treatment and are ineffective;
   3. Those who have relapsed within 12 months after CR after consolidation and intensive treatment;
   4. Those who relapse after 12 months but are ineffective after conventional chemotherapy;
   5. Subjects who experienced relapses twice or multiple times; with persistent extramedullary leukemia.
6. Kidney function, cardiopulmonary function, liver function, and coagulation function meet the following requirements:

   1. Creatinine ≤ 1.5 ULN;
   2. Left ventricular ejection fraction ≥ 50% and echocardiography does not reveal pericardial effusions and ECG does not reveal clinically significant abnormal bands;
   3. Blood oxygen saturation > 92%;
   4. Total bilirubin ≤ 2 × ULN; ALT and AST ≤ 2.5 × ULN; for the patients with ALT and AST abnormalities caused by disease which researchers judge (e.g. liver infiltrates or bile duct obstruction), the indicators of which can be relaxed to ≤5× ULN;
   5. PT/INR and PTT ≤ 1.5 ULN;
7. Patients understand the trial and have signed the informed consent form.

Exclusion Criteria:

1. Patients with malignant tumors other than acute myeloid leukemia within 5 years before the screening, except fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after the radical operation, and breast ductal carcinoma in situ after radical operation;
2. Patients with hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal reference range; Hepatitis C virus (HCV) antibody positive and hepatitis C virus (HCV) RNA positive in peripheral blood; Human immunodeficiency virus (HIV) antibody-positive; Cytomegalovirus (CMV) DNA positive; Syphilis test positive;
3. Patients with severe heart disease: including but not limited to unstable angina pectoris, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade III), severe arrhythmia;
4. Patients with unstable systemic diseases judged by the researcher: including but not limited to severe liver, kidney, or metabolic diseases requiring drug treatment;
5. Within 7 days before screening, there were active or uncontrollable infections requiring systemic treatment (except mild urogenital infection and upper respiratory tract infection);
6. Pregnant or lactating women, female subjects who planned pregnancy within 2 years after cell reinfusion, or male subjects whose partners planned pregnancy within 2 years after cell reinfusion;
7. Subjects who were receiving systemic steroid treatment within 7 days before screening or who were determined by the investigator to need long-term systemic steroid treatment during treatment (except inhalation or local use);
8. Participated in other clinical studies within 1 month before screening;
9. There was evidence of central nervous system invasion during subject screening(e.g. detection of tumor cells in cerebrospinal fluid or imaging suggests central infiltrates;);
10. Patients with graft-versus-host disease (GVHD) or requiring immunosuppressive agents;
11. Patients with a history of epilepsy or other central nervous system disorders;
12. Patients with primary immunodeficiency diseases;
13. Patients who are not suitable for cell construction judged by researchers;
14. Other situation researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerable dose (MTD) | within 2 yeas after infusion
  Fludarabine + Cyclophosphamide + TAA05 Cell Injection Patients will receive lymphodepletion with fludarabine (25 mg/kg) and cyclophosphamide (250 mg/kg) for 3 days on day -7~-2, followed by the infusion of TAA05 Cell with the dose of 1×10^8, 2×10^8 or 4×10^8 cells on day 0. If no dose-limited toxicity(DLT) emerges in the group, then the subsequent higher dose will be used in the next group. If DLT emerges in a single subject in any dose level, 3 more subjects will be enrolled to the same dose level. MTD is defined as the highest dose at which DLT occurs in no more than 2 of the 6 patients. After the end of dose climbing, if the maximum dose group(MTD) is still not observed, the highest dose group is defined as MTD.

SECONDARY OUTCOMES:
Incidence of Treatment-related Adverse Events | within 2 yeas after infusion
  Adverse events will be assessed according to NCI-CTCAE v5.0, cytokine release syndrome and CAR-T cell-related encephalopathy syndrome will be assessed according to ASTCT criteria.
Overall response rate(ORR) of administering Anti-FLT3 CAR-T Cell in Relapsed/Refractory Acute Myeloid Leukemia | within 2 yeas after infusion
  OR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Complete response rate(CRR) of administering Anti-FLT3 CAR-T Cell in Relapsed/Refractory Acute Myeloid Leukemia | within 2 yeas after infusion
  CRR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Overall survival(OS) of administering Anti-FLT3 CAR-T Cell in Relapsed/Refractory Acute Myeloid Leukemia | within 2 yeas after infusion
  OS will be assessed from CAR T cell infusion to death or last follow-up (censored).
Progress-free survival(PFS) of administering Anti-FLT3 CAR-T Cell in Relapsed/Refractory Acute Myeloid Leukemia | within 2 yeas after infusion
  PFS will be assessed from CAR T cell infusion to death or last follow-up (censored).
Duration of Response(DOR) of administering Anti-FLT3 CAR-T Cell in Relapsed/Refractory Acute Myeloid Leukemia | within 2 yeas after infusion
  DOR will be assessed from CAR T cell infusion to death or last follow-up (censored).
In vivo expansion and survival of Anti-FLT3 CAR-T Cell | within 2 yeas after infusion
  Quantity of CAR copies in bone marrow and peripheral blood will be determined by using qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen L, Mao H, Zhang J, Chu J, Devine S, Caligiuri MA, Yu J. Targeting FLT3 by chimeric antigen receptor T cells for the treatment of acute myeloid leukemia. Leukemia. 2017 Aug;31(8):1830-1834. doi: 10.1038/leu.2017.147. Epub 2017 May 12. No abstract available. PMID 28496177